CLINICAL TRIAL: NCT01257009
Title: Atorvastatin Reduces Sympathetic Activity in Patients With Chronic Kidney Disease
Brief Title: Atorvastatin and Sympathetic Activity in Chronic Kidney Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Statin sympathetic
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-11

CONDITIONS: Stable Chronic Kidney Disease; Hypertension
Keywords: sympathetic activity; chronic kidney disease; atorvastatin; lipitor
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Arm 1: cessation of any statin therapy for at least 6 weeks, then the first sympathetic activity measurement will be done.Subsequently, atorvastatin 20mg is added for 6 weeks. Then the second sympathetic measurement will be performed.
  Interventions: Drug: Atorvastatin
- 2 (Other): Patients will receive atorvastatin for 6 weeks, then the first sympathetic measurement will be done. Then atorvastatin will be stopped and 6 weeks the second measurement will be done
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — 6 weeks treatment with atorvastatin and studying the effect of atorvastatin on sympathetic activity
  Other Names: Lipitor

SUMMARY:
Hypertensive chronic kidney disease (CKD) patients often have sympathetic hyperactivity which appears to contribute to the pathogenesis of hypertension and cardiovascular organ damage. Experimental studies and some clinical studies have shown that statin therapy can reduce central sympathetic activity. Blockade of the renin-angiotensin system (RAS), which is standard treatment for CKD, is known to lower sympathetic activity.

The investigators hypothesize that adding a statin for 6 weeks to RAS blockade would further lower sympathetic activity in hypertensive stage 2-4 CKD patients.

Methods: In ten stable CKD patients who are on chronic treatment with renin-angiotenis blockers, blood pressure and sympathetic activity (quantified by assessment of muscle sympathetic nerve activity, MSNA) will be assessed at baseline and 6 weeks after atorvastatin 20mg/day added.

Ten other CKD patients will serve as time control and will be studied twice with an interval of 6 weeks without any change in medication, to quantify within subject reproducibility.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* stable chronic kidney disease
* Hypertension

Exclusion Criteria:

* renal replacement therapy
* pregnancy
* diabetes mellitus

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2009-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Sympathetic activity | 4-6 weeks treatment

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center utrecht, Utrecht, Utrecht, Netherlands